CLINICAL TRIAL: NCT04966832
Title: A Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics of XW10508 Immediate and Modified Release Formulations in Healthy Adults
Brief Title: Safety, Tolerability and Pharmacokinetics of XW10508 Immediate and Modified Release Formulations in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XWPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XW10508-101
Record Dates: First submitted 2021-07-12; First posted 2021-07-19 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: In this double-blind study, participants will be randomized to XW10508 or placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XW10508 (Experimental): XW10508 capsules or tablets
  Interventions: Drug: XW10508
- Placebo (Placebo Comparator): Placebo capsules or tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: XW10508 — XW10508 capsules or tablets
  Arms: XW10508
Other: Placebo — Placebo capsules or tablets
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of XW10508 in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-in-human single and multiple ascending oral dose pharmacokinetic and safety study where participants will receive either XW10508 or placebo. Both immediate release and modified release formulations will be assessed. Timed blood samples will be collected to assess the pharmacokinetics after the study drug is ingested by the participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants who are 18 to 55 years of age, inclusive.
* Participant is willing and able to provide signed and dated written informed consent to participate prior to admission to the study.

Exclusion Criteria:

* Evidence or history of clinically significant (in the opinion of the investigator) gastrointestinal, hepatic, renal, respiratory (e.g., asthma, COPD), cardiovascular (e.g., hypertension), metabolic, psychiatric, neurological, immunological, or endocrine disorders, or allergic disease including drug allergies, including immediate type hypersensitivity to components of the study drug. A history of childhood asthma that has resolved is acceptable.
* Use of tobacco- or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, patches, vaping device, etc.) within 3 months prior to Day -1 and/or positive urine cotinine test at Screening or Day -1.
* Participant who, for any reason, is deemed by the investigator to be inappropriate for this study; or has any condition which would confound or interfere with the evaluation of the safety, tolerability, pharmacokinetics or pharmacodynamics of the investigational drug; or is unable to comply with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and causality of adverse events (AEs) | Up to 12 Days

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | 48 hours
Trough concentration (Cmin) | 48 hours
Area under the concentration-time curve (AUC) from 0 to time of last quantifiable concentration | 48 hours
AUC from time 0 extrapolated to infinity (AUC0-inf) | 48 hours
AUC over the dosing interval (AUCtau) | 48 hours
Apparent terminal half-life (t1/2) | 48 hours
Cmax and AUC ratios of metabolites to XW10172 | 48 hours
Time to reach Cmax (Tmax) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Canafax, PharmD, Study Director — XWPharma
Locations (1):
- CMAX, Adelaide, South Australia, Australia